CLINICAL TRIAL: NCT00128713
Title: Determination of the Optimal Prophylactic Platelet Dose Strategy to Prevent Bleeding in Thrombocytopenic Patients (A TMH CTN Study)
Brief Title: Optimal Platelet Dose Strategy for Management of Thrombocytopenia
Acronym: PLADO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Transfusion Medicine/Hemostasis Clinical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 238; U01HL072268 (NIH); U01HL072028 (NIH); U01HL072033 (NIH); U01HL072072 (NIH); U01HL072191 (NIH); U01HL072196 (NIH); U01HL072248 (NIH); U01HL072274 (NIH); U01HL072283 (NIH); U01HL072289 (NIH); U01HL072290 (NIH); U01HL072291 (NIH); U01HL072305 (NIH); U01HL072331 (NIH); U01HL072346 (NIH); U01HL072355 (NIH); U01HL072359 (NIH)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2013-08

CONDITIONS: Thrombocytopenia
Keywords: Blood Transfusion; Blood Platelets
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Lower Dose Prophylactic Platelets
  Interventions: Procedure: Lower Dose Prophylactic Platelet Transfusions
- 2 (Active Comparator): Medium Dose Prophylactic Platelets
  Interventions: Procedure: Medium Dose Prophylactic Platelet Transfusions
- 3 (Active Comparator): Higher Dose Prophylactic Platelets
  Interventions: Procedure: Higher Dose Prophylactic Platelet Transfusions

INTERVENTIONS:
Procedure: Medium Dose Prophylactic Platelet Transfusions — 2.2 x 10^11 platelets per m^2 BSA
  Arms: 2
Procedure: Lower Dose Prophylactic Platelet Transfusions — 1.1 x 10^11 platelets per m^2 BSA
  Arms: 1
Procedure: Higher Dose Prophylactic Platelet Transfusions — 4.4 * 10^11 platelets per m^2 BSA
  Arms: 3

SUMMARY:
The primary objective of this study is to compare the three study arms of lower, medium, and higher dose platelet therapy with respect to the percentage of patients experiencing at least one episode of Grade 2 or higher bleeding as determined by the Platelet Dose Trial Bleeding Scale (Grade 2 bleeding corresponds to bleeding that is moderate, but not severe enough to warrant red blood cell transfusion).

There are a number of secondary endpoints related to platelet transfusions, hemostasis, and other concerns. The four most important secondary endpoints will compare the three study arms with respect to the following outcomes: 1) platelet utilization rates (total number of platelets transfused x 10 ^11); 2) number of platelet transfusion events (frequency of transfusions); a transfusion event would be defined as each separate platelet transfusion issued by the study site's transfusion service; 3) highest category of bleeding during time of study (Platelet Dose Trial Bleeding Scale Grades less than or equal to 1, 2, 3, or 4 by arm); and 4) bleeding severity based on number of days with bleeding (total days of bleeding and bleeding/thrombocytopenic day), intensity of bleeding, and number of sites with bleeding (if such a severity score has been validated and published by the time the study is completed).

DETAILED DESCRIPTION:
BACKGROUND:

It is important to identify the safest and most cost effective strategies for providing platelet support that will achieve effective disease management without depleting platelet supplies. Informative clinical data have been provided concerning the platelet transfusion trigger. In contrast, the optimal quantity of platelets to be used per transfusion remains a highly controversial subject. No prospective platelet transfusion studies have been performed in which patients are randomized to an assigned platelet dose throughout their period of thrombocytopenia.

DESIGN NARRATIVE:

After obtaining consent and verifying eligibility requirements, the patients will be randomized to one of three doses for prophylactic platelet transfusions (lower, medium, or higher dose). The dosage is based on the patient's body surface area (BSA). The dose targets are as follows: 1) the lower dose is 1.1 x 10^11/m²; 2) the medium dose is 2.2 x 10^11/m²; and 3) the higher dose is 4.4 x 10^11/m². A dose within 25% of this value in either direction is considered to be in the target range. For many adult patients, the typical dose of one unit of apheresis platelets would fall in the target range for the medium dose. All prophylactic transfusions provided while the patient is in the study will be given according to the randomized target dose range. Only blood bank staff, not clinical staff, will have access to the target dose range for each patient.

The patient's morning platelet count will be taken every day. If this value is less than or equal to 10,000, a prophylactic platelet transfusion will be given. Otherwise, no prophylactic platelet transfusion will be given that day. Platelet transfusions may be given at any time, and at any dose, to treat active bleeding or in association with an invasive procedure. A hemostatic assessment will be carried out every day to identify any bleeding the patient may experience. This assessment involves a patient interview, physical assessment, and a chart review. Data on all transfusions (e.g., platelets and red blood cells), all transfusion-related events, all serious adverse events, and protocol deviations will also be recorded.

Patients will participate in the study either until 30 days after the initial platelet transfusion, until they have not received a platelet transfusion for 10 days after the most recent platelet transfusion, or until hospital discharge (whichever comes first).

Each of the three pairwise dose comparisons is of interest. Therefore, the primary and secondary endpoints will be analyzed using three separate pairwise comparisons, each at the 0.017 significance level to adjust for multiple comparisons.

This study has been approved by the National Heart, Lung, and Blood Institute (NHLBI)-appointed protocol review committee and data and safety monitoring board (DSMB), and each participating institution's institutional review board. An interim monitoring plan was developed by the protocol team and DSMB, and is described in the protocol. The study is being monitored in accordance with this plan.

ELIGIBILITY:
Inclusion Criteria:

* Has, or is expected to have, hypoproliferative thrombocytopenia, and is expected to have a platelet count of up to 10,000 ul for at least 5 days and be in the hospital for at least 5 days
* Weight is between 10 and 135 kilograms
* PT/INR, PTT, and fibrinogen assays that are measured within 72 hours before study entry are as follows:

  1. PT less than or equal to 1.3 times the upper limit of normal for the laboratory
  2. PTT less than or equal to 1.3 times the upper limit of normal for the laboratory
  3. Fibrinogen greater than or equal to 100 mg/dl
* Undergoing, or has completed, hematopoietic stem cell transplantation, for any diagnosis; OR has a diagnosis of acute or chronic leukemia, non-Hodgkins or Hodgkins lymphoma, myeloma, myelodysplasia, or non-hematologic malignancy and is undergoing, or has completed, chemotherapy
* During this hospitalization, the patient has not yet received any platelet transfusions related to the current or planned course of therapy (individual platelet transfusions given prior to the study and unrelated to thrombocytopenia will not exclude the patient)

Exclusion Criteria:

* Evidence of greater than or equal to Grade 2 bleeding (as determined by the Platelet Dose Trial Bleeding Scale)
* Receiving antithrombotic drugs
* Will receive bedside leuko-reduced platelet transfusions
* Present, or history of, platelet transfusion refractoriness within 30 days prior to study entry
* Pre-enrollment lymphocytotoxic antibody screen (PRA) known to be greater than or equal to 20% based on prior data
* Present, or history of, acute promyelocytic leukemia (APML), immune thrombocytopenic purpura (ITP), thrombotic thrombocytopenic purpura (TTP), or hemolytic-uremic syndrome (HUS)
* Will be transfused at platelet trigger of greater than 10,000 platelets/ul
* Recent history of major surgery (within 2 weeks of study entry)
* Currently taking, or participating in a study involving, platelet substitutes, platelet growth factors, or pharmacologic agents intended to enhance or decrease platelet hemostatic function
* Pregnant
* Previously enrolled in this study

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F. Assmann, Principal Investigator — New England Research Institutes, Inc.; Mark Brecher, MD, Principal Investigator — University of North Carolina; James B. Bussel, MD, Principal Investigator — NY-Presbyterian Hosp/Weill Cornell Medical Center; James George, MD, Principal Investigator — U of Oklahoma Health Sciences Center; John R. Hess, Principal Investigator — University of Maryland, Baltimore; Christopher D. Hillyer, MD, Principal Investigator — Emory University; Barbara A. Konkle, MD, Principal Investigator — University of Pennsylvania; Cindy A. Leissinger, MD, Principal Investigator — Tulane University; Keith R. McCrae, MD, Principal Investigator — University Hospitals Cleveland; Jeffrey McCullough, MD, Study Chair — University of Minnesota; Janice G. McFarland, MD, Principal Investigator — Versiti Blood Health; Paul M. Ness, MD, Principal Investigator — Johns Hopkins University; Ellis Neufeld, MD, PhD, Principal Investigator — Boston Children's Hospital; Thomas L. Ortel, MD, PhD, Principal Investigator — Duke University; Sherrill J. Slichter, MD, Study Chair — Bloodworks; Ronald G. Strauss, MD, Principal Investigator — University of Iowa; Darrell J. Triulzi, MD, Principal Investigator — University of Pittsburgh Presbyterian and Shadyside Hospital
Locations (21):
- United States (21):
  - Emory University Hospitals; Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Tulane University Hospital and Clinics, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston; Beth Israel Deaconess Medical Center; Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - NY-Presbyterian Hosp/Weill Cornell Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital Cleveland, Cleveland, Ohio
  - U of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - U of Pennsylvania Health System; Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian and Shadyside Hospital, Pittsburgh, Pennsylvania
  - U of Texas SW Medical Center at Dallas, Dallas, Texas
  - Virginia Mason Hospital, Seattle, Washington
  - U of Washington Medical Center/FHCRC; Children's Hospital and Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Oncology Alliance/St. Luke's Hospital, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Uhl L, Assmann SF, Hamza TH, Harrison RW, Gernsheimer T, Slichter SJ. Laboratory predictors of bleeding and the effect of platelet and RBC transfusions on bleeding outcomes in the PLADO trial. Blood. 2017 Sep 7;130(10):1247-1258. doi: 10.1182/blood-2017-01-757930. Epub 2017 Jul 5. PMID 28679741
- [Derived] Josephson CD, Granger S, Assmann SF, Castillejo MI, Strauss RG, Slichter SJ, Steiner ME, Journeycake JM, Thornburg CD, Bussel J, Grabowski EF, Neufeld EJ, Savage W, Sloan SR. Bleeding risks are higher in children versus adults given prophylactic platelet transfusions for treatment-induced hypoproliferative thrombocytopenia. Blood. 2012 Jul 26;120(4):748-60. doi: 10.1182/blood-2011-11-389569. Epub 2012 Apr 26. PMID 22538854
- [Derived] Triulzi DJ, Assmann SF, Strauss RG, Ness PM, Hess JR, Kaufman RM, Granger S, Slichter SJ. The impact of platelet transfusion characteristics on posttransfusion platelet increments and clinical bleeding in patients with hypoproliferative thrombocytopenia. Blood. 2012 Jun 7;119(23):5553-62. doi: 10.1182/blood-2011-11-393165. Epub 2012 Apr 10. PMID 22496156
- [Derived] Slichter SJ, Kaufman RM, Assmann SF, McCullough J, Triulzi DJ, Strauss RG, Gernsheimer TB, Ness PM, Brecher ME, Josephson CD, Konkle BA, Woodson RD, Ortel TL, Hillyer CD, Skerrett DL, McCrae KR, Sloan SR, Uhl L, George JN, Aquino VM, Manno CS, McFarland JG, Hess JR, Leissinger C, Granger S. Dose of prophylactic platelet transfusions and prevention of hemorrhage. N Engl J Med. 2010 Feb 18;362(7):600-13. doi: 10.1056/NEJMoa0904084. PMID 20164484

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower Dose Platelets: Lower Dose Prophylactic Platelets (1.1 x 10^11 per m^2 Body Surface Area per transfusion, +/- 25%)
- Medium Dose Platelets: Medium Dose Prophylactic Platelets (2.2 x 10^11 per m^2 Body Surface Area per transfusion, +/- 25%)
- Higher Dose Platelets: Higher Dose Prophylactic Platelets (4.4 x 10^11 per m^2 Body Surface Area per transfusion, +/- 25%)
Period: Overall Study
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Started | 453 | 449 | 449
Completed | 453 | 449 | 449
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets | Total
Number analyzed (Participants) | 453 | 449 | 449 | 1351
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (19.3) | 44.7 (19.3) | 45.5 (19.7) | 44.6 (19.4)
Age, Customized [Number; unit: participants]
  0 - 17 years | 67 | 68 | 64 | 199
  18 - 20 years | 9 | 6 | 8 | 23
  >=21 years | 377 | 374 | 377 | 1128
  Unknown/not reported | 0 | 1 | 0 | 1
Sex/Gender, Customized [Number; unit: participants]
  Female | 189 | 176 | 169 | 534
  Male | 264 | 272 | 280 | 816
  Unknown/not reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 3 | 8
  Asian | 7 | 8 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Black or African American | 53 | 37 | 40 | 130
  White | 362 | 374 | 378 | 1114
  More than one race | 13 | 9 | 10 | 32
  Unknown or Not Reported | 12 | 20 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 21 | 58
  Not Hispanic or Latino | 433 | 425 | 423 | 1281
  Unknown or Not Reported | 2 | 5 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 453 | 449 | 449 | 1351
Treatment Regimen [Number; unit: Participants]
  Autologous or syngeneic stem cell transplant | 154 | 149 | 151 | 454
  Allogeneic stem cell transplant | 185 | 185 | 186 | 556
  Chemotherapy for hematologic malignancy | 111 | 112 | 110 | 333
  Chemotherapy for solid tumor | 3 | 3 | 2 | 8
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.8 (0.4) | 1.8 (0.4) | 1.8 (0.4) | 1.8 (0.4)
Height [Mean (Standard Deviation); unit: cm] | 165.5 (21.4) | 164.0 (21.7) | 166.2 (19.3) | 165.2 (20.8)
Weight [Mean (Standard Deviation); unit: kg] | 77.4 (24.9) | 75.0 (26.3) | 76.0 (23.8) | 76.1 (25.0)

OUTCOME MEASURES:

1. Primary Outcome: At Least One Day With Grade 2 or Higher Bleeding
Description: Any Grade 2 (moderate) or higher grade bleeding, as determined by daily hemostatic assessment and documentation of any red blood cell transfusions to treat bleeding
Time Frame: From randomization until the subject ends the study (10 days after most recent platelet transfusion, 30 days after first platelet transfusion on study, or hospital discharge, whichever occurs first)
Population: These analyses were done on an intention-to-treat basis. That is, patients were counted in the treatment arm to which they were randomly assigned, even if they actually received transfusions that were not according to their assigned dosing strategy.
Measure: Number; unit: participants
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Number analyzed (Participants) | 446 | 435 | 434
participants
  Yes | 304 | 293 | 299
  No | 142 | 142 | 135
  Not Evaluable | 7 | 14 | 15
Statistical Analysis 1: Comparison: Lower Dose Platelets vs Medium Dose Platelets; Test type: Superiority or Other; p = 0.83, Fisher Exact — Three one-degree-of-freedom chi-square tests, each comparing a pair of treatment groups. These tests were carried out at the .017 significance level to adjust for the multiple comparisons; These tests were carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 2: Comparison: Lower Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p = 0.83, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; These tests were carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 3: Comparison: Medium Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p = 0.66, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; These tests were carried out at the .017 significance level to adjust for the multiple comparisons

2. Secondary Outcome: Platelet Utilization
Description: Total number of platelets transfused, based on attempted dose, among subjects who have at least one platelet transfusion and no missing data on attempted doses.
Time Frame: as for outcome 1
Population: Subjects with missing information and those that did not receive at least one platelet transfusion were excluded from the analysis.
Measure: Median (Full Range); unit: Number of platelets (x10^11)
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Number analyzed (Participants) | 357 | 387 | 395
Number of platelets (x10^11) | 10.96 [0.67 to 196.35] | 12.49 [1.06 to 487.33] | 22.43 [2.49 to 363.66]
Statistical Analysis 1: Comparison: Lower Dose Platelets vs Medium Dose Platelets; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney) — All analyses are based on intention to treat. These tests were carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 2: Comparison: Lower Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Medium Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Platelet Transfusion Episodes
Description: Number of platelet transfusion episodes among subjects who have at least one platelet transfusion and no missing data on attempted doses.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Number of platelet transfusion episodes
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Number analyzed (Participants) | 357 | 387 | 395
Number of platelet transfusion episodes | 5 [1 to 58] | 3 [1 to 111] | 3 [1 to 44]
Statistical Analysis 1: Comparison: Lower Dose Platelets vs Medium Dose Platelets; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — All analyses were carried out using intention to treat. These tests were carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 2: Comparison: Lower Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Medium Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Bleeding Severity, if a Suitable Scale is Validated and Published by the Time the Trial Ends
Description: No suitable scale was identified, so no analyses for this outcome were carried out
Time Frame: as for outcome 1
Population: Analysis not performed; no applicable bleeding severity scale validated and published by end of PLADO Study
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Highest Grade of Bleeding While on Study
Description: Highest grade of bleeding during time on study using Platelet Dose Trial modification of World Health Organization Bleeding Scale. Grades 0-1 (no or minimal bleeding), 2 (moderate bleeding), 3 (bleeding generally requiring red cell transfusion), 4 (severe bleeding)
Time Frame: as for outcome 1
Population: The analysis was done as intention to treat. Subjects for which highest grade of bleeding could not be determined (non-evaluable) were excluded.
Measure: Number; unit: participants
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Number analyzed (Participants) | 435 | 423 | 424
participants
  Grade 0 or 1 (no bleeding or minimal bleeding) | 142 | 142 | 135
  Grade 2 (moderate bleeding) | 245 | 244 | 249
  Grade 3 (bleeding generally requiring RBC's) | 36 | 27 | 33
  Grade 4 (severe bleeding) | 12 | 10 | 7
  Not Evaluable | 18 | 26 | 25
Statistical Analysis 1: Comparison: Lower Dose Platelets vs Medium Dose Platelets; Test type: Superiority or Other; p = 0.51, Mantel Haenszel — Each pair of treatment arms was compared using an exact version of the Mantel-Haenszel test for trend; These tests will be carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 2: Comparison: Lower Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p = 0.82, Mantel Haenszel — Each pair of treatment arms was compared using an exact version of the Mantel-Haenszel test for trend; These tests will be carried out at the .017 significance level to adjust for the multiple comparisons
Statistical Analysis 3: Comparison: Medium Dose Platelets vs Higher Dose Platelets; Test type: Superiority or Other; p = 0.68, Mantel Haenszel — Each pair of treatment arms was compared using an exact version of the Mantel-Haenszel test for trend; These tests will be carried out at the .017 significance level to adjust for the multiple comparisons

ADVERSE EVENTS:
Time Frame: For serious adverse events (SAE): from randomization until the subject ends the study. For adverse events (AE) other than SAEs: during and within the 4 hours following each transfusion.
Description: Subjects ended the study 10 days after most recent platelet transfusion, 30 days after first platelet transfusion on study, or at hospital discharge or death, whichever occurs first.
  Throughout their time on study, subjects were hospitalized. Assessment for AE and SAE was through review of medical records and daily assessment of subject.
Arm/Group | Lower Dose Platelets | Medium Dose Platelets | Higher Dose Platelets
Serious Adverse Events (participants affected / at risk) | 38/453 | 27/449 | 36/449
Other Adverse Events (participants affected / at risk) | 197/453 | 182/449 | 203/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Platelets (N=453) | Medium Dose Platelets (N=449) | Higher Dose Platelets (N=449)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Angioedema and Mucositis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrilation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain - Probably Due To Chemotherapy Toxicity (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Colonic Ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 4 (5) | 0 (0) | 0 (0)
Failed Engraftment (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever with Hypoxia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever, Rigors and Shortness of Breath (General disorders) | 0 (0) | 0 (0) | 1 (1)
Graft-Versus-Host Disease (Immune system disorders) | 0 (0) | 0 (0) | 3 (3)
Heart Block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hemodynamic Instability (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hemoptysis and Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (General disorders) | 1 (1) | 0 (0) | 2 (2)
Hypotension and Possible Sepsis (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension and Hypoxemia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension and Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intracranial Bleed (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intubation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ischemia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Multisystem Organ Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Obtunded Level of Consciousness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Perforated Appendix (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (1)
Possible Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Possible Toxoplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Relapse of Acute Myelogenous Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 7 (7)
Respiratory Distress and Multiorgan Failure (General disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Distress and Renal Failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1)
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 3 (3) | 5 (5)
Sepsis and Multiorgan Failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Septic Shock and Renal Failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subdural Hematoma (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Transfusion Related Acute Lung Injury vs Fluid Overload (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Veno-Occlusive Disease (Hepatobiliary disorders) | 6 (6) | 5 (5) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Platelets (N=453) | Medium Dose Platelets (N=449) | Higher Dose Platelets (N=449)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 37 (50) | 46 (60) | 55 (82)
Sinus Bradycardia (Cardiac disorders) | 4 (6) | 5 (6) | 6 (7)
Sinus Tachycardia (Cardiac disorders) | 43 (91) | 41 (86) | 35 (54)
Hypertension (General disorders) | 39 (81) | 34 (61) | 46 (75)
Hypotension (General disorders) | 32 (52) | 23 (28) | 25 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 20 (30) | 18 (22)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 15 (19) | 14 (18)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (3) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 7 (8)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (3)
Rigors, chills (General disorders) | 37 (55) | 42 (55) | 49 (72)
Fever (General disorders) | 153 (425) | 133 (333) | 143 (358)
Infection (Infections and infestations) | 4 (6) | 4 (4) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No